CLINICAL TRIAL: NCT04480788
Title: Early Clinical Study on Increasing Dose and Open Label of T Cell Injection Targeting CD7 Autologous Chimeric Antigen Receptor in the Treatment of Relapsed / Refractory CD7 Positive Hemolymph System Malignancies
Brief Title: CD7-CART in the Treatment of r / r CD7 Positive Hemolymph System Malignancies on Increasing Dose and Open Label Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-CART-07-001
Record Dates: First submitted 2020-07-14; First posted 2020-07-21 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: T Lymphoblastic Leukemia/Lymphoma; Extramedullary NK-T-cell Lymphoma, Nasal Type; Peripheral T-cell Lymphoma, Nonspecific; Angioimmunoblastic T-cell Lymphoma; Enteropathy-Associated T-Cell Lymphoma; Anaplastic Large Cell Lymphoma, ALK-negative; T-cell Lymphoblastic Leukemia
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Peripheral; Immunoblastic Lymphadenopathy; Enteropathy-Associated T-Cell Lymphoma; Lymphoma, Large-Cell, Anaplastic

STUDY DESIGN:
Intervention Model Description: CD7-CART
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- T cell injection targeting CD7 chimeric antigen receptor (Experimental)
  Interventions: Biological: T cell injection targeting CD7 chimeric antigen receptor

INTERVENTIONS:
Biological: T cell injection targeting CD7 chimeric antigen receptor — Drug name: T cell injection targeting CD7 autologous chimeric antigen receptor. Package specification: 10-50ml bag, 1-4 bags / person, which is determined according to the body weight of the subject and the effective content of cell preparation

SUMMARY:
Phase I was a single arm, open label, dose increasing study to explore the safety, tolerance and Cytodynamic characteristics of the drug, and to preliminarily observe the efficacy of the study drug in relapsed / refractory CD7 Positive hematolymph system malignant tumor patients, so as to explore the clinical applicable dose of phase II. Since the activity and toxicity of cellular drugs (long-term survival drugs) do not have obvious dose dependence, and the increase of their dose may be accompanied by the increase of toxicity, rather than necessary for therapeutic effect, it is not necessarily suitable to recommend the effective dose according to the maximum tolerable dose (MTD). Therefore, this study will be based on the safety data, as well as the preliminary efficacy, efficacy and drug The end point of pharmacokinetics (ORR, the content of CD7 Positive Cells, the expansion and duration of car-t cells) were comprehensively considered to determine the recommended dose for phase II clinical trial.Main research purposes Objective to evaluate the safety and tolerability of T cell injection targeting CD7 autologous chimeric antigen receptor in the treatment of relapsed / refractory CD7 Positive hematological and lymphoid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* The age ranged from 7 to 70 years (including the cut-off value), regardless of gender
* The expected survival time was more than 6 weeks
* ECOG score 0-1
* Malignant lymphoma (including but not limited to acute T-lymphoblastic leukemia / lymphoma; extramedullary NK / T-cell lymphoma, nasal type; peripheral T-cell lymphoma, nonspecific; vascular immunoblastic T-cell lymphoma; intestinal disease associated T-cell lymphomas; anaplastic large cell lymphoma (ALK -); T-cell lymphoblastic leukemia)
* When screening, hematological malignancies with CD7 Positive confirmed by bone marrow examination or tumor pathology with positive rate of CD7 ≥ 30%, meeting one of the following conditions:

  1. At least two chemotherapy regimens failed or did not achieve complete remission or relapse;
  2. Patients who relapsed after stem cell transplantation were not affected by other treatment methods;
* For peripheral blood involved acute T-lymphoblastic leukemia / lymphoma and NK / T-cell lymphoma, patients with TCR rearrangement were detected by ngs
* The liver and kidney function, heart and lung function meet the following requirements:

  1. Creatinine ≤ 1.5 ULN;
  2. LVEF ≥ 45%;
  3. Blood oxygen saturation > 91%;
  4. The total bilirubin ≤ 2 × ULN; ALT and AST ≤ 2.5 × ULN; the abnormal ALT and AST caused by diseases (such as liver infiltration or bile duct obstruction) can be relaxed to ≤ 5 × ULN;
* Understand the experiment and have signed the informed consent

Exclusion Criteria:

* Those who need immunosuppressant;
* For intestinal disease-related T-cell lymphoma, patients with intestinal ulcer or hematochezia were examined by colonoscopy;
* In addition to cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical operation, and breast ductal carcinoma in situ after radical operation;
* The patients with positive HBsAg or HBcAb and HBV DNA titer in peripheral blood were not within the normal reference value; those with positive anti HCV antibody and positive HCV RNA in peripheral blood; those with HIV antibody positive and cytomegalovirus DNA positive Syphilis was positive;
* Severe heart disease: including but not limited to unstable angina pectoris, myocardial infarction (within 6 months before screening), congestive heart failure (NYHA classification ≥ III), severe arrhythmia;
* Unstable systemic diseases judged by researchers: including but not limited to severe liver, kidney or metabolic diseases requiring drug treatment;
* Within 7 days before screening, there were active or uncontrollable infections requiring systemic treatment (except for mild genitourinary system infection and upper respiratory tract infection);
* Pregnant or lactating women, female subjects planning pregnancy within 1 year after cell reinfusion or male subjects whose partners plan to conceive within 1 year after cell reinfusion;
* Patients who had received car-t therapy or other gene modified cell therapy before screening;
* Subjects who were receiving systemic steroid therapy or were receiving systemic steroid therapy for 7 days were excluded;
* Participated in other clinical studies within 3 months before screening;
* There was evidence of central nervous system invasion during screening;
* According to the judgment of the researchers, it does not conform to the condition of cell preparation;
* Other researchers think it is not suitable to be included in the study.

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 2 years

SECONDARY OUTCOMES:
Safety results | Up to 2 years
  Number of adverse events
PK | Up to 2 years
  The maximum concentration (Cmax）
PK | Up to 2 years
  the time to reach the maximum concentration (Tmax)
PK | Up to 2 years
  The area under the curve (auc0-28d ) at 28d respectively after administration
PD | Up to 2 years
  Absolute value of CD7 Positive Cells in peripheral blood at each time point
PD | Up to 2 years
  The proportion of CD7 Positive Cells in peripheral blood at each time point
ORR | Up to 2 years
  The total response rate was 3 months and 6 months
overall survival (OS) | Up to 2 years
  Time from initiation of CD7 car-t cell therapy to death (for any reason)
Search Results Featured snippet from the web Duration of response (DOR) | Up to 2 years
  The time from the first assessment of Cr or PR to the first assessment of recurrence or progression of the disease or death from any cause
Progression-free survival (PFS) | Up to 2 years
  The time from the beginning of treatment with CD7 car-t cells to the first progression of disease or death from any cause
Immunogenicity | Up to 2 years
  The positive rate of human anti car antibody at each time point

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China